CLINICAL TRIAL: NCT06161129
Title: Filter Lenses for the Prevention of Migraine Attacks - Effects of Blue Cut and FL-41 Filter Lenses
Brief Title: Filter Lenses for the Prevention of Migraine Attacks
Acronym: COMFORT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rune Skovgaard Rasmussen (Other)
Collaborators: Center of Communication (CSU-Slagelse) (Unknown)
Responsible Party: Sponsor-Investigator, Rune Skovgaard Rasmussen, Associate professor of pathology, neuropsychologist, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 108314
Record Dates: First submitted 2023-11-16; First posted 2023-12-07 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Migraine; Glasses; Headache; Visual Impairment
Keywords: Migraine; filter glasses; pain; headache; treatment
MeSH Terms: conditions — Migraine Disorders; Headache; Vision Disorders; Pain | interventions — Lenses

STUDY DESIGN:
Intervention Model Description: Four arms will be used:
  1: Control. 2. BlueCut filter. 3. FL-41 filter. 4. Below 500 nm filter.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not meet each other. Outcome assessors and participants will not know which type of filters are used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control (No Intervention): Group of 50 participants (control) will receive glasses with clear lenses.
- FL-41 (Active Comparator): Group of 50 participants will receive a glasses with an FL-41 filter.
  Interventions: Device: Lenses
- BlueCut (Active Comparator): Group of 50 participants will receive glasses with a Blue Cut filter.
  Interventions: Device: Lenses
- 500nm (Active Comparator): Group of 50 participants will receive glasses with a below 500 nm filter
  Interventions: Device: Lenses

INTERVENTIONS:
Device: Lenses — The filter lenses will be worn by participants for one month all day.
  Arms: 500nm; BlueCut; FL-41

SUMMARY:
The purpose is to investigate whether the Blue Cut for Night filter is better at reducing migraine compared to the FL-41 filter or a filter blocking light below 500 nm. A control group will use clear lenses without filter. This is a controlled, randomized and double-blind trial.

DETAILED DESCRIPTION:
Migraine is a neurological disorder that often causes severe, throbbing headaches that can be accompanied by nausea and vomiting. In addition, sound or light sensitivity is often seen. An attack can last up to 72 hours. Migraine can occur in one half of the head and is exacerbated by physical activity. There are several different types of migraine, of which the inherited migraine typically cannot be cured. Migraine affects about 15% of all adults worldwide, but about twice as many women as men.

About 10% of diagnosed patients have chronic migraine, which is characterized by at least 15 days of severe headache each month. Many patients have tension headaches between attacks.

Migraine most often starts in the most productive years of life, between the ages of 20 and 50, and most affects the age group of 35-54 years. For many women, migraine debuts after childbirth, while others experience that it disappears after childbirth. Several women experience that they get migraine when they have their period. This migraine is called hormonal and can follow them for many years.

Several studies have shown that migraine attacks are triggered by light, and many become very light-sensitive during an attack. So far, a FL 41 lens, which excludes blue-green light, has been the only migraine-specific optical treatment.

A new lens called "Blue Cut for Night Glass" has in a study resulted in participants experiencing less migraine. For 4 weeks, 10 participants used only the lens in the evening. Results showed that they had fewer days with headaches. The lens is so new that it has not yet come into regular production and trade. In connection with the present study, the investigators have received 13 sets of lenses.

For many years, FL-41 has been the preferred filter lens for the prevention of migraine attacks, since it was first successfully tested on children in 1991. Since this study, much has happened in terms of the development of filter lenses.

The purpose is to investigate whether the Blue Cut for Night filter is better at reducing migraine compared to the FL-41 filter or a filter blocking light below 500 nm. A control group will use clear lenses without filter. This is a controlled, randomized and double-blind trial.

ELIGIBILITY:
Inclusion criteria:

* Adult individuals below the age of 66.
* Diagnosed with migraine by a neurologist.
* Able to communicate in Danish
* Able to voluntarily come to the clinic during an untreated migraine attack.
* Must have had migraine attacks for more than 1 year.

Exclusion criteria:

* Fewer than four migraine attacks per month.
* Chronic neck pain
* Chronic headache
* Chronic use of opioids
* Presence of a pathological eye condition (in the study, an eye condition is defined as a permanent eye condition that affects the front and back of the eye, such as glaucoma, age-related macular degeneration)
* Other acquired and congenital retinal diseases must not be present.
* If there is more than 1 line of deviation on the Snellen chart from habitual correction to best correction, the participant must have a new pair of glasses made at their own expense.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Change of pain intensity during migraine attacks | Measured at inclusion, 4 weeks after inclusion, and 8 weeks after inclusion
  Intensity is described from 1-10 on a visual analog pain scale (VAS). A score of 1 is very mild intensity and 10 is very severe.

SECONDARY OUTCOMES:
Headache Impact Test (HIT-6) | Measured at inclusion, 4 weeks after inclusion, and 8 weeks after inclusion
  Headache Impact Test (HIT-6), which is a validated questionnaire. It consists of 6 questions and assesses participants' functional status in the past 4 weeks. The questions measure the frequency and severity of headaches, as well as their consequences for the participant's activity level. The scale scores from 36 to 78, with a high score being the worst. This questionnaire is recommended by the Danish Medicines Council for Danish migraine patients
Migraine-Specific Quality-of-Life Questionnaire v. 2.1 (MSQ) | Measured at inclusion, 4 weeks after inclusion, and 8 weeks after inclusion
  MSQ is a frequently used disease-specific survey for assessing health-related quality of life in people with migraine. MSQ is validated for persons with episodic migraine and persons with chronic migraine. MSQ measures quality of life within the last 4 weeks in relation to restrictive function, preventive function, and emotional function. The score ranges from 0-100, with a higher score indicating improvement in quality of life
Monthly migraine days | Every day of participation lasting 8 weeks
  The date of the migraine attack, duration, and medication used are noted. A migraine day is defined as a day on which the person experienced a migraine attack or used medication to relieve acute attacks
Fatigue Severity Scale | Measured at inclusion, 4 weeks after inclusion, and 8 weeks after inclusion
  Short fatigue questionnaire used to assess the occurrence of disabling fatigue. There are 9 items scored from 1 to 7, where 7 indicated the most fatigue. A score of 63 is worst, and disabling fatigue may be observed scoring 45 or more points.
Groffman Visual Tracing Test | Measured at inclusion, 4 weeks after inclusion, and 8 weeks after inclusion
  Test for assessment of attention, visuospatial function, and figure-ground perception. The test is stressful and requires a high degree of sustained visual focus, and can be expected to be affected by pain, fatigue, light sensitivity, and oculomotor dysfunction
The Migraine Disability Assessment Test | Measured at inclusion, 4 weeks after inclusion, and 8 weeks after inclusion
  The questionnaire is changed to a 1-month focus period instead of 3 months. The Migraine Disability Assessment Test is frequently used to measure the effectiveness of interventions for migraine
Medication use, both as needed (PN) and daily fixed medication | Every day of participation lasting 8 weeks
  Consumption of preparations and dosage is recorded in a diary
Major Depression Inventory | Measured at inclusion, 4 weeks after inclusion, and 8 weeks after inclusion
  About 80% of people with chronic migraine are affected by depression. Major Depression Inventory is used in the present study to monitor for symptoms of depression as well as part of the assessment of mental well-being and quality of life
The 36-Item Health Survey | Measured at inclusion, 4 weeks after inclusion, and 8 weeks after inclusion
  The 36-Item Health Survey is used to measure quality of life and is frequently used to measure the effectiveness of different treatments for headache-affected persons. The questionnaire has 8 dimensions ranging for 0 to 100 points, where a high score indicates better functioning. The 8 dimensions are: physical functioning, role physical, bodily pain, general health perceptions, vitality, social function, role emotional, og mental health.
Assessment of photophobia via questionnaire | Measured at inclusion, 4 weeks after inclusion, and 8 weeks after inclusion
  Assessment of photophobia via questionnaire, where each participant assesses their own light sensitivity during the day, at night, and indoors. This is done both with and without filter glasses. The amount of photophobia is measured on a scale from 0 to 10, where 10 indicates maximum and worst photophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Smaakjær, MSc, Principal Investigator — CSU-Slagelse
Locations (1):
- CSU-Slagelse, Slagelse, Denmark

IPD SHARING:
Plan to Share IPD: No